CLINICAL TRIAL: NCT04857099
Title: Retrospective Study Within the Brugmann University Hospital of the Navilas ® Micropulse Laser Treatment for Macular Edema
Brief Title: Impact of the Navilas ® Micropulse Laser Treatment for Macular Edema Within the CHU Brugmann Hospital Macular Edema
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Laurence Postelmans, Head of the Ophtalmology Department, Brugmann University Hospital
Other Study IDs: CHUB-Kemani
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Macular edema
  Interventions: Other: Data extraction from medical files

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
The Navilas® micropulse laser can be used to treat patients with macular edema and good visual acuity, which therefore do not fall within the indications for conventional treatments by intravitreal injections.

The CHU Brugmann Hospital is the only center to own this laser in Belgium.This study aims to evaluate the efficacy of this laser.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse macular edema without focal edema source accessible by focal laser (e.g. capillary telangiectasia)
* Central retinal thickness ≤ 400microns.
* Patient does not meet the reimbursement criteria for intra-vitreous injections(IVI) of anti-VEGF (eg AV> 5/10).
* IVI are contraindicated.
* Physician considers that it is preferable to space out the injections because of the side effects (eg. ocular disturbance during IVI, eye pain, sensation of a foreign body, spots in the visual field generating a visual gene etc.)
* Patient wishing to space the anti-VEGF IVI.

Exclusion Criteria:

* Macular edema of a different etiology than diabetic macular edema or venous thrombosis (e.g. cataract extraction, vitreomacular traction, epiretinal membrane etc.)
* Central retinal thickness > 400 microns.
* The eye presents a focal edematous maculopathy accessible to conventional laser.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective study including 23 files of patients treated with the Navilas ® micropulse laser, in the period from 04/25/2018 to 11/10/2020
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Baseline versus three months after treatment
Retinal thickness change | Baseline versus three months after treatment
Periodicity of anti-VEGF injections | Baseline versus three months after treatment
Scar - assessed by optical coherence tomography | Three months after treatment
Scar - assessed by fluorescein angiography | Three months after treatment
Scar - assessed by auto-fluorescence fundus images | Three months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roman Kemani, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No